CLINICAL TRIAL: NCT01299922
Title: Phase III, Open, Randomized, Parallel-group Clinical Trial, to Evaluate the Efficacy and Safety of Treatment With Prednisone, Cyclosporine, Mycophenolic Acid Versus Prednisone and Mycophenolic Acid in Lupus Nephritis Type III-IV-V.
Brief Title: Clinical Trial Treatment in Lupus Nephritis
Acronym: Csa-LES
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: IT was impossible to find patients
Sponsor: Hospital Universitario Fundación Alcorcón (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Infanta Sofia (Other); Hospital Universitario Infanta Leonor (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital Regional Universitario Carlos Haya (Other); Hospital Universitario Virgen de la Victoria (Other); University Hospital of the Nuestra Señora de Candelaria (Other); Hospital Universitario de Guadalajara. Spain (Unknown); Hospital San Pedro de Alcantara (Other); Hospital Juan Canalejo (Other)
Responsible Party: Manuel Praga Terente, Hospital Universitario Doce de Octubre Madrid Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Csa-LES
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2011-02

CONDITIONS: Lupus Nephritis
Keywords: Lupus nephritis; Therapy; Cyclosporin; Mycophenolic acid
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cyclosporine+mycophenolic acid+prednison (Experimental): Triple therapy
  Interventions: Drug: cyclosporine +mycophenolic acid+prednison
- mycophenolic acid + prednison (Active Comparator): Mycophenolic acid+prednison 106 weeks
  Interventions: Drug: Mycophenolic Acid + prednison

INTERVENTIONS:
Drug: cyclosporine +mycophenolic acid+prednison — Cyclosporine for 26 weeks Prednisone+mycophenolic acid 106 weeks
  Other Names: Triple therapy
  Arms: cyclosporine+mycophenolic acid+prednison
Drug: Mycophenolic Acid + prednison — Mycophenolic Acid + prednison for 106 weeks
  Other Names: Conventional therapy
  Arms: mycophenolic acid + prednison

SUMMARY:
The treatment of lupus nephritis with cyclophosphamide and steroids changed the prognosis of lupus nephritis in the early '80s. In recent years, alternative regimens have appeared in both the induction and maintenance with similar results at least to those offered by the classic pattern and possibly with fewer side effects, especially for long term. The association of prednison and mycophenolate has created large expectations to that effect, and is part of first-line therapeutic arsenal of lupus nephritis type III, IV and V.

Despite the significant advances that have led to these treatments, the likelihood of complete remission after six months remains, according to the series of 8-13% and partial remission do not exceed 60% in papers published. In the last year, two articles have been published supporting the use of triple therapy (prednisone, mycophenolate, cyclosporine) in poor prognosis of lupus nephritis with hopefully better results than those obtained previously. In this study we try to compare the effectiveness of triple therapy, the therapy is now considered standard (prednisone, mycophenolate) in patients with lupus nephritis type III-IV-V

DETAILED DESCRIPTION:
asd

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients diagnosed SLE with renal type III-IV-V confirmed by renal biopsy done in the last 6 months
* Proteinuria > 2 g/24 hours and hematuria (> 5 h / field)
* MDRD4 eGFR > 60 ml/min/1.73m2
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Central nervous system LES involvement or any other vital organ
* Active infection
* Use of mycophenolic acid, mycophenolate mofetil, cyclosporine or tacrolimus in the last 6 months
* No adherence
* Women of childbearing age not using appropriate contraceptive methods.
* Positive pregnancy test
* Anasarca
* Malignancy or cancer history (except basal cell skin carcinomas)
* Patient participating in another study with an investigational drug or have participated within 28 days prior to entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
the number of complete remissions, between the triple therapy with cyclosporine-prednisone-mycophenolic acid and conventional therapy with mycophenolic acid-prednisone as induction therapy in patients with lupus nephritis type III-IV-V | 36 months
  Complete remission:
  * Proteinuria < 0.3 g/24h
  * Albumin normal
  * eGFR > 60 mL/min/1.73 m2

SECONDARY OUTCOMES:
the number of partial and complete remissions, between triple therapy with prednisone, cyclosporine, mycophenolic acid and prednisone-mycophenolic acid. | 36 months
  Partial remission: Proteinuria 0.3-3.5 g/24 hours, with a decrease > 50% over basal, stable renal function and albumin normal
the number of patients with adverse effects | 36 months
the rate (%) of decline of proteinuria in two groups | 36 months
the decrease in GFR (ml/min/1.73m2) in both groups | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernandez Juarez Gema, MD Ph, Study Director — Hospital Universitario Fundación Alcorcón; Praga Terente Manuel, MD Ph, Study Chair — Hospital Universitario Doce de Octubre
Locations (1):
- Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid, Spain